CLINICAL TRIAL: NCT01681641
Title: Managing Changes in Life After Deep Brain Stimulation for Parkinson's Disease - Designing and Developing a Targeted Nursing Program to Patients and Spouses.
Brief Title: Managing Changes in Life After Deep Brain Stimulation for Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AUHN-0211-AH
Record Dates: First submitted 2012-08-13; First posted 2012-09-10 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2012-09

CONDITIONS: Parkinson's Disease
Keywords: Patients; Nursing; Parkinsons disease; Deep Brain Stimulation; Spouses
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Experimental): Patients and spouses in the intervention group are offered 3 targeted meetings with the DBS nurse, focusing on goal setting for each individual, following DBS, based on patients and spouses own expectations, challenges and goals for everyday life after DBS.
  Interventions: Other: A psycho-social intervention
- Control group (No Intervention): Patients and spouses enrolled in a control group

INTERVENTIONS:
Other: A psycho-social intervention
  Arms: Lifestyle counseling

SUMMARY:
Parkinson's disease is a chronic progressive neurological disorder. Symptoms are tremor, slowness in movement, rigidity and postural instability. As the disease progresses and treatment with L-dopa is no longer sufficient, some patients may be treated with deep brain stimulation.

When treated with deep brain stimulation, electrodes are inserted in the affected area of the brain and through stimulation, motor symptoms of Parkinson's disease are significantly reduced.

During the first year of DBS treatment patients and spouses may experience changes in everyday life and illness trajectory posing new opportunities as well as new challenges.

The purpose of the study is to develop an individualised and targeted nursing program to support patients and relatives manage changes and challenges in life the first three months after Deep Brain Stimulation. The intervention is expected to generate important knowledge that will serve as a foundation for the further development of a future nursing program.

DETAILED DESCRIPTION:
The intervention is designed as a psychosocial intervention, targeted both patients and spouses.

The intervention consists of individually targeted meetings with a specialized DBS nurse several times during the first six months og DBS. Patients and spouses likewise have to fill out a diary for use in the meetings.

All meetings have specific topics, addressing aspects of challenges in adjusting to DBS, and the aim is to off patients and spouses a tailored intervention, supporting each individual based on an individual assessment.

ELIGIBILITY:
Inclusion Criteria:

* eligible and offered treatment with DBS for PD
* married or cohabitant

Exclusion Criteria:

* living alone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in sense of Coherence in intervention group compared to control group | Baseline, 6 months, 12 months
  Questionnaire

SECONDARY OUTCOMES:
Quality of life | Baseline, 6 months, 12 months
  PDQ 39 or PDQ Carer

OTHER OUTCOMES:
Qualitative interviews | 12 months
  Patients and spouses experience of participating in the intervention. Perceived use of knowledge gained

CONTACTS AND LOCATIONS:
Overall Officials: Anita Haahr, PHD, Principal Investigator — Department of Neurology, Aarhus University Hospital
Locations (3):
- Denmark (3):
  - Department of Neurology, Aarhus University Hospital, Aarhus, Jutland
  - Department of Neurology , Aarhus University Hospital, Aarhus
  - Bispebjerg Hospital, Copenhagen

IPD SHARING:
Plan to Share IPD: No